CLINICAL TRIAL: NCT01343537
Title: Real Time Continuous Neurophysiological Monitoring for Early Detection of Cerebral Vasospasm in Aneurysmal Subarachnoid Hemorrhage Subjects
Brief Title: Continuous Neurophysiological Monitoring Detection of Cerebral Vasospasm in Aneurysmal Subarachnoid Hemorrhage Subjects
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5981
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2011-04

CONDITIONS: Cerebral Vasospasm; SAH; Aneurysm
Keywords: Brain Bleed; SAH; Vasospasm
MeSH Terms: conditions — Vasospasm, Intracranial; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Monitoring (Experimental)
  Interventions: Other: Neuro Monitoring

INTERVENTIONS:
Other: Neuro Monitoring — Neuro monitoring from day 4 to day 14 post subarachnoid hemorrhage for cerebral vasospasm

SUMMARY:
Aneurysmal subarachnoid hemorrhage (bleeding on the brain due to a ruptured aneurysm) is a serious condition with a high morbidity (incidence of having ill health) and mortality (death). There are approximately 11 cases per 100,000 in the population per year, and approximately 40% of these cases are fatal. (Ingall) Among the fortunate subjects who survive the initial bleed, vasospasm and subsequent stroke are a major cause of morbidity. Vasospasm is defined as a prolonged severe, although reversible cause of arterial narrowing that occurs after bleeding into the subarachnoid space, most commonly after aneurysmal rupture. (Youman) The reduced arterial diameter inhibits blood flow and deprives the brain of oxygen, which often results in a stroke.

Vasospasm is a major problem when treating subjects with aneurysmal subarachnoid hemorrhage. For these reasons, it is essential to diagnose cerebral vasospasm early, before permanent deficits develop.

There may be another option to solve this dilemma. The field of neuro-monitoring (neurological monitoring) has the technology available to continuously monitor brain activity of these sedated ICU subjects. This may allow for early diagnosis and possibly identify changes in neurologic function before they become symptomatic. In the past, neuro-monitoring was primarily used in the operating room to monitor neurologic function during surgery in and around the spinal cord. Surgery to the spine or spinal cord also carries its own form of risk, either from mechanical trauma to the spinal cord or its nerve roots, or from interruption of the blood supply to these structures. Should damage to nerve fibers occur, the end result could be paralysis, loss of sensation, and onset of severe burning (i.e. neuropathic) pain. The field of intraoperative neuro-monitoring (IOM) was developed to address these risks during spine surgery, whereby nerves rostral (toward the head) or caudal (toward the feet) to the site of surgery are stimulated (usually via electrical pulses) and signals are recorded from the side opposite to the site of stimulation. Thus, the signals carried by nerve fibers are forced to pass through the region at risk from the surgery. In the event that changes in nerve responses are seen, the surgical team is notified, and they can change what they're doing to try and restore signals, thereby preserving function in the nerve fibers.

This same technology has been used in the neurosurgical ICU to monitor subjects with severe brain injury from trauma, stroke, intracranial hemorrhage and subarachnoid hemorrhage. Using continuous electroencephalogram (EEG) monitoring combined with somatosensory evoked potentials (SSEPs) (a type of neuro monitoring) has been used to determine prognosis, identify subjects in subclinical status epilepticus (state of brain being in a constant seizure), predict elevations in the intracranial pressure Increased pressure within the skull), and diagnose cerebral hypoxia (not enough oxygen in the brain) (Amantini)

DETAILED DESCRIPTION:
Aneurysmal subarachnoid hemorrhage is a serious condition with a high morbidity and mortality. There are approximately 11 cases per 100,000 population per year, and approximately 40% of these cases are fatal. (Ingall) Among the fortunate subjects who survive the initial bleed, vasospasm and subsequent stroke are a major cause of morbidity. Vasospasm is defined as a prolonged severe, although reversible cause of arterial narrowing that occurs after bleeding into the subarachnoid space, most commonly after aneurismal rupture. (Youman) The reduced arterial diameter inhibits blood flow and deprives the brain of oxygen, which often results in a stroke.

Vasospasm is a major problem when treating subjects with aneurismal subarachnoid hemorrhage. Up to 75% of subjects with aneurismal subarachnoid hemorrhage will develop vasospasm, and 30% of subarachnoid hemorrhage subjects will become clinically symptomatic, with muscle weakness as the primary symptom. (Dorsch) Even with intervention, 12% of patents with symptomatic vasospasm will develop permanent clinical deficits (after a ruptured aneurysm) including hemiplegia, aphasias, and visual loss. Less severe strokes may lead to modest loss of strength and sensation on one side of the body, and/or deterioration in higher brain functions, such as memory, speech comprehension, and planning.

Continuous Neuro-monitoring has previously been used in the trauma ICU setting as a means to detect deterioration in brain function after closed head injury (Amantini, Daubin), ischemic encephalopathy (Hakimi) and in subjects with MCA stroke to determine function (Tzvetanov). It was also observed that monitoring changes occur prior to ICP elevations in critically ill subjects (Amantini). These studies have demonstrated the feasibility as well as the safety of monitoring in an ICU.

No studies to date have attempted monitoring for vasospasm in subjects who suffered an aneurysmal subarachnoid hemorrhage. Motor evoked potential have also not been trialed in the ICU, although MEP may be more useful to determine both cerebral ischemia, as well as functional outcome.

ELIGIBILITY:
All adult subjects who have a subarachnoid hemorrhage from a ruptured aneurysm and require high levels of sedation, or a poor neurologic exam and mechanical ventilation will be eligible for the study. Hunt and Hess Grade 4 and 5(worst grades; highest mortality; highest level of dependence if survived) subarachnoid hemorrhage subjects by definition have a severely depressed exam, and will require intubation and mechanical ventilation. Those subjects whose respiratory status deteriorates necessitating intubation and high levels of sedation will also qualify.

All subjects who have subarachnoid hemorrhage from undetermined source, such as angiogram negative subarachnoid hemorrhage, those who have a reliable neurological exam such as Hunt and Hess grade 1-3 subarachnoid hemorrhage subjects, and those who are intubated, but require minimal sedation and therefore have a consistent neurological exam will be excluded from the study. Also, any subject that has a body temperature of less then 32 degrees Celsius will be excluded.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Early detection of cerebral vasospasm after aneurysmal subarachnoid hemorrhage | One year
  To determine the feasibility and safety using intermittent motor evoked potentials, somatosensory evoked potentials and EEG monitoring to detect vasospasm compared against our standard detection methods including transcranial doppler ultrasound, computed tomography angiogram, computed tomography perfusion scan and the gold standard: formal cerebral angiography

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Deshaies, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States